CLINICAL TRIAL: NCT03390114
Title: Internet-Based Cognitive Behavioral Therapy to Treat Insomnia in HIV: A Pilot Trial
Brief Title: Cognitive Behavioral Therapy to Treat Insomnia in Persons With HIV Infection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Samir K Gupta, MD, MS, Professor of Medicine, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1712469162
Record Dates: First submitted 2017-12-28; First posted 2018-01-04 (Actual); Results first posted 2021-02-21 (Actual); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: HIV/AIDS; Insomnia
Keywords: HIV; Insomnia; Cognitive Behavioral Therapy
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: 10-week, randomized, controlled, single-blinded, two-arm, parallel group, pilot trial at a single center
Who Masked: Investigator
Masking Description: The primary investigator is blinded to the treatment assignment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SHUTi Cognitive Behavioral Therapy (Experimental): SHUTi (www.myshuti.com) is an evidence-based, cognitive-behavioral, online intervention for insomnia.
  Interventions: Behavioral: SHUTi
- Usual Care (No Intervention): Patients randomized to the Usual Care group will be encouraged to follow-up with their primary care or HIV provider. There will be no formal interaction with the participants between the Entry Visit and the Week 10 Visit. However, the participants will be encouraged to contact the study team for any changes in their condition. There will be no restrictions on the care that can be received, although we will assess changes in care during the trial.

INTERVENTIONS:
Behavioral: SHUTi — SHUTi consists of six, 40-minute, weekly sessions during which the intervention components of stimulus control, sleep restriction, sleep hygiene, cognitive restructuring, and relapse prevention are delivered. Each SHUTi session has the same structure: the main content, a homework screen with options, and a summary of the main points.
  Arms: SHUTi Cognitive Behavioral Therapy

SUMMARY:
The goal of this preliminary study is to determine the efficacy of an internet-based treatment program for insomnia for HIV-infected persons.

DETAILED DESCRIPTION:
The primary objective of this pilot trial is to compare 10-week changes in Insomnia Severity Index (ISI) scores in HIV-infected adults with clinically relevant insomnia severity and who are already receiving virologically suppressive antiretroviral therapy (ART) and are then randomized to either treatment with the SHUTi cognitive behavioral therapy program or to Usual Care (UC). A total of 100 persons with HIV may be screened to identify the 32 participants to be enrolled and randomized into the pilot trial. These participants will be ≥ 18 years old, have been receiving antiretroviral therapy with an HIV viral load < 75 copies/mL within three months of the Entry Visit, and have an ISI score ≥ 15 within three months of the Entry Visit. These participants will be randomized 1:1 (stratified by age <40 vs. ≥ 40 years) to either insomnia treatment with the SHUTi cognitive behavioral therapy program (N=16) or usual care (N=16).

ELIGIBILITY:
Inclusion Criteria:

1. HIV-1 infection, documented by both: (1) any licensed rapid HIV test or HIV enzyme test kit at any time prior to study entry and (2) by at least one detectable HIV-1 antigen or at least one detectable plasma HIV-1 RNA viral load.
2. Age equal to or greater than 18 years.
3. Ongoing receipt of antiretroviral therapy of any kind for at least 3 months prior to the Entry Visit.
4. HIV-1 RNA level < 75 copies/mL obtained during routine clinical care within 90 days of the Entry Visit.

   NOTE: There are no CD4 cell count eligibility criteria for this trial.
5. ISI score ≥ 15

Exclusion Criteria:

1. Inability to complete written, informed consent.
2. Incarceration at the time of any study visit.
3. Active suicidality, as determined by the patient's HIV provider or social worker following a positive response (1, 2, or 3) to PHQ-9 Item #9
4. Diagnosed vascular disease (documented history of angina pectoris, coronary disease, peripheral vascular disease, cerebrovascular disease, aortic aneurysm, or otherwise known atherosclerotic disease).
5. History of congestive heart failure, even if currently compensated.
6. Diagnosed disease or process, besides HIV infection, associated with increased systemic inflammation (including, but not limited to, systemic lupus erythematosis, inflammatory bowel diseases, other collagen vascular diseases).

   Note: Hepatitis B or C co-infections are NOT exclusionary
7. Known or suspected malignancy requiring systemic treatment within 180 days of the Entry Visit.

   NOTE: Localized treatment for skin cancers is not exclusionary.
8. Uncontrolled hyperthyroidism or hypothyroidism, defined as TSH values outside of the local reference range on most recent clinical assessment.
9. Last known clinic-based estimated glomerular filtration rate (eGFR) < 50 mL/min/1.73m2. (calculated from the 2009 CKD-EPI equation).
10. Uncontrolled diabetes defined as the last known clinic-based Hgb A1C > 8.0 g/dL.
11. Last known clinic-based total cholesterol > 240 mg/dL.
12. Therapy for serious medical illnesses within 14 days prior to screening.

    Note: Therapy for serious medical illnesses that overlaps with a main study visit will result in postponement of that study visit until the course of therapy is completed; postponement outside of the allowed study visit timeframe will result in study discontinuation.
13. Pregnancy or breastfeeding during the course of the study.
14. Receipt of investigational agents, cytotoxic chemotherapy, systemic glucocorticoids (of any dose), or anabolic steroids at the Entry Visit.

    Note: Physiologic testosterone replacement therapy or topical steroids is not exclusionary. Inhaled/nasal steroids are not exclusionary as long as the participant is not also receiving HIV protease inhibitors.
15. Active drug use or dependence that, in the opinion of the investigator, would interfere with adherence to study requirements.
16. History of schizophrenia, bipolar disorder, or dementia.

    NOTE: Depression is not exclusionary as long as the severity of depression does impede ability to perform the required study procedures.
17. Musculoskeletal or neurologic disorders that impede ability to perform the required study procedures.
18. History of sleep apnea or restless leg syndrome.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Samir K Gupta, MD, MS, Principal Investigator — Indiana University School of Medicine
Locations (1):
- Infectious Diseases Research Center, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be made available to other researchers. These include demographics, medical history/medication history, ISI scores, and changes in ISI scores by study arm.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: Data will become available within 30 days of completion of final statistical analysis. There is no expiration of data availability.
Access Criteria: Please contact the study PI, Dr. Samir Gupta, for specific details on data availability.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | SHUTi Cognitive Behavioral Therapy | Usual Care
Started | 10 | 10
Completed | 6 | 8
Not Completed | 4 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SHUTi Cognitive Behavioral Therapy | Usual Care | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.2 (11.4) | 47.0 (14.7) | 46.6 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 8 | 9 | 17
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 9 | 8 | 17
  White | 1 | 1 | 2
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Insomnia Severity Index
Description: Change in the Insomnia Severity Index (ISI) score as measured by questionnaire. The ISI score ranges from 0 to 28 with higher scores indicating greater severity in insomnia symptoms.
Time Frame: 10 weeks
Population: Those who completed both pre and post assessments
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SHUTi Cognitive Behavioral Therapy | Usual Care
Number analyzed (Participants) | 6 | 8
score on a scale | -9.0 (9.4) | -3.4 (2.0)

ADVERSE EVENTS:
Time Frame: 10 weeks
Arm/Group | SHUTi Cognitive Behavioral Therapy | Usual Care
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Informed Consent Form (2018-11-09): https://cdn.clinicaltrials.gov/large-docs/14/NCT03390114/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2019-02-13): https://cdn.clinicaltrials.gov/large-docs/14/NCT03390114/Prot_SAP_001.pdf